CLINICAL TRIAL: NCT04332549
Title: A Randomized, Open Label, Two Period, Single Dose, Crossover, Bioavailability Study of Paclitaxel Injection Concentrate for Suspension (PICS) in Subjects With Locally Recurrent or Metastatic Breast Cancer.
Brief Title: To Assess the Bioavailability and Safety of Paclitaxel Injection Concentrate for Suspension in Subjects With Locally Recurrent or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: After meeting with the FDA, SPARC concludes a BE study will not be required
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SDO-006-20-01
Record Dates: First submitted 2020-03-26; First posted 2020-04-02 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Metastatic Breast Cancer; Locally Recurrent Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Reconstitution Method 1 (Active Comparator)
  Interventions: Drug: PICS (Reconstitution Method 1 or 2)
- Reconstitution Method 2 (Active Comparator)
  Interventions: Drug: PICS (Reconstitution Method 1 or 2)

INTERVENTIONS:
Drug: PICS (Reconstitution Method 1 or 2) — dose: 260mg/m2 Frequency: 2 period cross over study Route of administration : intravenous infusion duration of therapy: 2 cycles of PICS

SUMMARY:
A randomized, multi center, open label, two-period, single dose, crossover study to evaluate the bioavailability and safety of Paclitaxel Injection Concentrate for Suspension in Locally Recurrent or Metastatic Breast Cancer subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has given written, informed consent (or legally acceptable representative /impartial witness when applicable) and is available for the duration of study
2. Histologically or cytologically confirmed diagnosis of breast cancer with adequate documentation of prior therapy with an anthracycline unless clinically contraindicated
3. Locally recurrent or MBC for which taxane-based therapy is an appropriate treatment option
4. Male or female aged greater than equal to 18 years
5. ECOG performance status less than equal to 1
6. Estimated life expectancy of at least 12 weeks
7. Adequate organ and immune system function as indicated by the following laboratory values, obtained less than equal to 2 weeks prior to dosing for Period 1 and Period 2:
8. Any chemotherapy, targeted therapy, major surgery, or irradiation must have been completed at least 4 weeks before enrollment (6 weeks for mitomycin C or nitrosurea); immune therapy or hormonal therapy (except palliative bisphosphonate therapy for bone pain) must be completed 2 weeks before enrollment and subjects must have recovered from all toxicities incurred as a result of previous therapy except alopecia; use of targeted therapy or antibody therapy should have been completed for at least 5 half-lives of the respective therapy before enrollment. Use of narcotic analgesics such as dihydrocodeine and medicinal herbs such as St. John's Wort, which may act as inhibitors/inducers of CYP2C8 and CYP3A4, must have been discontinued at least 2 weeks and 4 weeks respectively before enrollment
9. Subjects of child bearing potential must practice an acceptable method of birth control as judged by the investigator

   * Medically acceptable methods of birth control include the use of either a contraceptive implant or a contraceptive injection (e.g., Depo-Provera™) or an intrauterine device, same sex partner or vasectomized partner or an oral contraceptive taken continually within the past three months and which the subject agrees to continue using during the study
   * To adopt another birth control method, or a double-barrier method which consists of a combination of any two of the following:

   diaphragm, cervical cap, condom, or a spermicide at least 2 months prior to study entry and must continue to use contraception for the duration of the study
10. Female subjects who are postmenopausal for at least 1 year as per investigator's discretion, or who are surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)
11. Male subjects enrolled in the trial cannot father a child and are advised to prevent passage of semen to their sexual partner during intercourse using acceptable methods as judged by the investigator for the duration of the study
12. Females subjects of child-bearing potential must have a negative urine pregnancy test
13. Female subjects must be non-lactating and non-breastfeeding
14. Subject must be willing and able to comply with scheduled visits, treatment plan and laboratory testing.

Exclusion Criteria:

1. Known hypersensitivity to the study drug or their excipients (cholesteryl sulfate, caprylic acid, polyvinylpyrrolidone, ethanol, polyethylene glycol)
2. Inability to undergo venipuncture and/or tolerate venous access
3. Presence of clinically symptomatic active CNS metastases, including leptomeningial involvement, requiring steroid or radiation therapy
4. Pre-existing clinically significant peripheral neuropathy (Grade 2 or higher according to CTCAE, Version 5.0)
5. Any other severe concurrent disease which in the judgment of the investigator would make the subject inappropriate for entry into this study or confound the study
6. Presence of pleural/ascitic fluid which cannot be definitively treated prior to dosing and during the PK blood draws in each period (Period 1 and Period 2) and if there is re-accumulation of fluid (greater than 5%) greater than 2 weeks after definitive management
7. Positive laboratory exclusion test (HIV, HBsAg, or HCV)
8. Treatment with investigational agents or participation in a clinical trial within 30 days of study entry
9. Failure of prior taxane therapy for metastatic disease or for adjuvant therapy within previous 6 months of screening visit
10. Subjects taking concurrent medications that may act as inhibitors/inducers of CYP2C8 and CYP3A4 within 2 weeks of screening and during Periods 1 and 2
11. Evidence or history of bleeding diathesis or coagulopathy within 6 months prior to screening visit
12. Uncontrolled cardiac disease, including: congestive heart failure (CHF) > Class II per New York Heart Association (NYHA), history of hypertensive crisis
13. Active clinical infection which in the treating investigator's opinion renders the subject ineligible or can confound the study
14. Serious non-healing wound, ulcer or bone fracture
15. Unresolved toxicity higher than CTCAE Version 5.0 Grade 1 (excluding alopecia, anemia) attributed to any prior therapy/procedure
16. History of gastrointestinal perforation within 6 months prior to screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-27 (Estimated); Primary Completion 2021-01-28 (Estimated); Study Completion 2021-01-28 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration Plasma | 8 weeks
area under the plasma concentration versus time curve, from time 0 to the last measurable concentration | 8 weeks
area under the plasma concentration versus time curve from time 0 to infinity | 8 weeks
Incidence of Treatment-Emergent Adverse Events | 8 weeks
  shall be coded per CTCAE, Version 5.0

CONTACTS AND LOCATIONS:
Locations (22):
- India (22):
  - SPARC Site 12, Visakhapatnam, Andhra Pradesh
  - SPARC Site 21, Ahmedabad, Gujarat
  - SPARC Site 22, Surat, Gujarat
  - SPARC Site 4, Bangalore, Karnataka
  - SPARC Site 10, Bangalore, Karnataka
  - SPARC Site 18, Bangalore, Karnataka
  - SPARC Site 13, Bangalore, Karnataka
  - SPARC Site 9, Aurangabad, Maharashtra
  - SPARC Site 8, Kolhāpur, Maharashtra
  - SPARC Site 2, Nagpur, Maharashtra
  - SPARC Site 1, Nagpur, Maharashtra
  - SPARC Site 17, Nagpur, Maharashtra
  - SPARC Site 3, Nashik, Maharashtra
  - SPARC Site 19, Nashik, Maharashtra
  - SPARC Site 15, Pune, Maharashtra
  - SPARC Site 16, Pune, Maharashtra
  - SPARC Site 5, Pune, Maharashtra
  - SPARC Site 11, Sangli, Maharashtra
  - SPARC Site 20, Khordha, Odisha
  - SPARC Site 14, Madurai, Tamil Nadu
  - SPARC Site 7, Lucknow, Uttar Pradesh
  - SPARC Site 6, Gujrāt, Vadodara

IPD SHARING:
Plan to Share IPD: No